CLINICAL TRIAL: NCT01963078
Title: Sex/Gender Differences in Risk and Resilience to PTSD; Implication of Oxytocin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Megan Moran-Santa Maria (Other)
Responsible Party: Sponsor-Investigator, Megan Moran-Santa Maria, Assistant Professor, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1R21MH099619-01 (NIH)
Record Dates: First submitted 2012-10-22; First posted 2013-10-16 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PTSD placebo Day 1, Oxytocin Day 2 (Placebo Comparator): Participants PTSD will self-administer matching placebo (containing all ingredients except OT) at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Interventions: Drug: Placebo
- PTSD Oxytocin Day 1, Placebo Day 2 (Experimental): Participants with PTSD will self-administer 24 IUs of OT nasal spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Interventions: Drug: Oxytocin
- Resilient Placebo Day 1, Oxytocin Day 2 (Placebo Comparator): Resilient controls will self-administer matching placebo spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Interventions: Drug: Placebo
- Resilient Oxytocin Day 1, Placebo Day 2 (Experimental): Resilient controls will self-administer 24 IUs of OT nasal spray at 10:30 a.m.on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Pitocin
  Arms: PTSD Oxytocin Day 1, Placebo Day 2; Resilient Oxytocin Day 1, Placebo Day 2
Drug: Placebo
  Other Names: Saline
  Arms: PTSD placebo Day 1, Oxytocin Day 2; Resilient Placebo Day 1, Oxytocin Day 2

SUMMARY:
The purpose of the study is to use fMRI to investigate amygdala response to fearful faces in men and women with and without PTSD who have experienced childhood trauma. The study will also compare the effects of oxytocin and placebo on amygdala response, and explore the interaction of oxytocin plasma levels and amygdala response in men and women with and without PTSD who have experienced childhood trauma.

Hypothesis 1: Amygdala responding will be greater in subjects with PTSD as compared to resilient subjects, and no sex differences in the magnitude of the response will be found.

Hypothesis 2A: In response to OT, women will exhibit a greater reduction in amygdala responding than men.

Hypothesis 2B: In response to OT, women with PTSD will exhibit a greater reduction in amygdala responding compared to women without PTSD.

Hypothesis 3A: Women with PTSD will have lower levels of plasma OT as compared to men with PTSD, and women and men without PTSD.

Hypothesis 3B: Plasma OT levels will be inversely correlated with amygdala responding to fearful faces in women but not in men.

ELIGIBILITY:
Inclusion Criteria

1. Ages 18-60.
2. Subjects scoring moderate to severe (>3) on a minimum of one of the five trauma domains of the Childhood Trauma Questionnaire.
3. Subjects must have experienced, witnessed, or confronted an event(s) that involved actual or threatened death or serious injury, or a threat to the physical integrity of themselves, or others and the person's response involved intense fear, helplessness, and/or horror (Criterion A DSM-IV for PTSD), prior to the age of 18.

Exclusion Criteria

1. Subjects with evidence of or a history of head trauma, neurological disorders, seizures, unconsciousness or any other major medical disorder.
2. Subjects with current (past 90 days) psychotic disorder or bipolar affective disorder.
3. Subjects with any psychoactive substance abuse within the last 30 days as evidenced by subject report or urine drug screen.
4. Women who are pregnant or nursing.
5. Women who are post-menopausal or have had a full hysterectomy.
6. Subjects who have a BMI greater than 35.
7. Subjects who are unwilling to maintain abstinence from alcohol and caffeine for the 24-hour period prior to the study visits and from illicit drug use for the 72 hour period prior to study visits.
8. Persons with ferrous metal implants or pacemaker.
9. Subjects who are claustrophobic.
10. Subjects taking endocrine or cardiovascular medications (other than blood pressure medications) during the 30-day period prior to the study.
11. Subjects with a postive breathalyzer or urine drug screen. Group - Specific Inclusion/Exclusion Criteria Individuals with PTSD Inclusion Criteria

1. Subjects must meet DSM-IV criteria for current (i.e. last 6 months) PTSD. 2. Subjects may also meet criteria for a mood disorder (except bipolar affective disorder, see Exclusion Criteria) or other anxiety disorders (panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder) or past (>90 days) alcohol dependence. The inclusion of subjects with affective and other anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with PTSD (Brady, Killeen, Brewerton, & Lucerini, 2000; Kessler, Chiu, Demler, Merikangas, & Walters, 2005).

Exclusion Criteria

1. As above.
2. Substance dependence within the past year, except for nicotine or alcohol. Resilient Controls Inclusion Criteria

1. As above. Exclusion Criteria

1. Subjects meeting criteria for current or past (i.e. last 90 days) Axis I mood or anxiety disorders (including PTSD and depression).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Moran- Santa Maria, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Clinical Neurosciences Division-Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Sippel LM, Flanagan JC, Holtzheimer PE, Moran-Santa-Maria MM, Brady KT, Joseph JE. Effects of intranasal oxytocin on threat- and reward-related functional connectivity in men and women with and without childhood abuse-related PTSD. Psychiatry Res Neuroimaging. 2021 Nov 30;317:111368. doi: 10.1016/j.pscychresns.2021.111368. Epub 2021 Aug 20. PMID 34455213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited primarily through media advertisements and flyers.
Groups:
- PTSD Placebo Day 1, Oxytocin Day 2: Participants PTSD will self-administer matching placebo (containing all ingredients except OT) at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Placebo
- PTSD Oxytocin Day 1, Placebo Day 2: Participants with PTSD will self-administer 24 IUs of OT nasal spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Oxytocin
- Resilient Placebo Day 1, Oxytocin Day 2: Resilient controls will self-administer matching placebo spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Placebo
- Resilient Oxytocin Day 1, Placebo Day 2: Resilient controls will self-administer 24 IUs of OT nasal spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Oxytocin
Period: Overall Study
Arm/Group | PTSD Placebo Day 1, Oxytocin Day 2 | PTSD Oxytocin Day 1, Placebo Day 2 | Resilient Placebo Day 1, Oxytocin Day 2 | Resilient Oxytocin Day 1, Placebo Day 2
Started | 9 | 10 | 10 | 9
Completed | 8 | 9 | 9 | 7
Not Completed | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Placebo Day 1, Oxytocin Day 2 | PTSD Oxytocin Day 1, Placebo Day 2 | Resilient Placebo Day 1, Oxytocin Day 2 | Resilient Oxytocin Day 1, Placebo Day 2 | Total
Number analyzed (Participants) | 9 | 10 | 10 | 9 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 10 | 9 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 7 | 22
  Male | 4 | 5 | 5 | 2 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 3 | 11
  White | 6 | 7 | 8 | 5 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Count of Participants]
  United States | 9 | 10 | 10 | 9 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Amygdala Activation- Oxy Minus Placebo
Description: Bold signal response to facial recognition task was contrasted between oxytocin and saline administrations. Participants with PTSD and Resilient Controls each underwent 2 sets of scanning procedures, one with placebo and one with Oxytocin. Participants were randomly assigned to received Oxytocin on Day 1 or Day 2, and placebo on the opposite day, to mitigate crossover effects. Outcome measure is change in bold signal response between the two days; bold signal response on placebo was subtracted from bold signal response on Oxytocin to obtain change score.
Time Frame: Days 1 and 2
Population: Population analyzed are participants who completed both scans and had usable MRI data.
Measure: Mean (Standard Deviation); unit: percentage of BOLD signal change
Arm/Group | PTSD Placebo Day 1, Oxytocin Day 2 | PTSD Oxytocin Day 1, Placebo Day 2 | Resilient Placebo Day 1, Oxytocin Day 2 | Resilient Oxytocin Day 1, Placebo Day 2
Number analyzed (Participants) | 8 | 9 | 9 | 7
percentage of BOLD signal change | -0.01 (0.36) | -0.02 (0.41) | 0.05 (0.54) | 0.21 (0.33)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant under both conditions, placebo and Oxytocin. Adverse events are reported summarily for each group.
Groups:
- PTSD Placebo: Participants PTSD will self-administer matching placebo (containing all ingredients except OT) at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Placebo
- PTSD Oxytocin: Participants with PTSD will self-administer 24 IUs of OT nasal spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Oxytocin
- Resilient Placebo: Resilient controls will self-administer matching placebo spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Placebo
- Resilient Oxytocin: Resilient controls will self-administer 24 IUs of OT nasal spray at 10:30 a.m. on Day 1 of study procedures, approximately 45-minutes prior the scanning sessions. This dose and timing of administration were selected based on similar fMRI studies (Domes, et al., 2007; Domes, et al., 2010; Kirsch, et al., 2005).
  Oxytocin
Arm/Group | PTSD Placebo | PTSD Oxytocin | Resilient Placebo | Resilient Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes